CLINICAL TRIAL: NCT04101578
Title: Prospective Observational Trial to Evaluate Clinical Prognosis and the Risk Factors for Progression for Myasthenia Gravis Patients
Brief Title: Clinical Prognosis and Progression of Myasthenia Gravis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Da, Yuwei, M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: 2017YFC0907705
Record Dates: First submitted 2019-09-16; First posted 2019-09-24 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Steroids; Immunosuppressive Agents; Immunoglobulins, Intravenous; Pyridostigmine Bromide; Prednisone; Methylprednisolone; Azathioprine; Tacrolimus; Cyclosporine; Cyclophosphamide; Mycophenolic Acid; Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples are collected annually.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ocular MG: Patients with autoimmune MG whose symptoms restricted to extraocular muscles
  Interventions: Drug: Symptomatic Treatment, Steroids, Immunosuppressive Agents, Plasma Exchange(PE), Intravenous Immunoglobulin(IVIg)
- Generalized MG: Patients not only suffer from extraocular muscles weakness but also from limb weakness, bulbar symptoms, or even respiratory failure
  Interventions: Drug: Symptomatic Treatment, Steroids, Immunosuppressive Agents, Plasma Exchange(PE), Intravenous Immunoglobulin(IVIg)

INTERVENTIONS:
Drug: Symptomatic Treatment, Steroids, Immunosuppressive Agents, Plasma Exchange(PE), Intravenous Immunoglobulin(IVIg) — Treatment regimens are determined according to the physician's judgment and preferences of the patients.
  Other Names: Pyridostigmine Bromide, Prednisone, Methylprednisolone, Azathioprine, Tacrolimus, Cyclosporin A, Cyclophosphamide, Mycophenolate Mofetil, Methotrexate

SUMMARY:
This study collects the clinical data of myasthenia gravis (MG) patients, assesses outcomes and adverse effects of different treatment regimens, and searches for risk factors of conversion to generalized MG.

DETAILED DESCRIPTION:
This is a multicenter, observational cohort trial in the real-world clinical setting recruiting MG patients from Neurology Departments of 6 hospitals in different regions of China. Clinical manifestations, laboratory test results, chest imaging and history of thymectomy are recorded. Patients will be classified by clinical manifestation as well as antibody status, and treatment regimens are determined according to the physician's judgment and preferences of the patients. Patients are followed up prospectively on regular to assess the outcomes of treatments and monitor any side effects. Peripheral blood samples are collected annually. Patients' clinical records are uploaded to an online database. The investigators plan to recruit a final sample of 2000 patients for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age >14.
2. Clinical Diagnosis of MG with supporting evidence:

   1. unequivocal clinical response to pyridostigmine
   2. positive antibody testing
   3. decrement >10% in repetitive nerve stimulations study (RNS) .
3. Willingness to sample collection, imaging study and other disease-related examinations and assessments.
4. Patients with informed consent.

Exclusion Criteria:

1. History of chronic degenerative, psychiatric, or neurologic disorder other than MG that can produce weakness or fatigue.
2. Age ≤14 years.
3. Severe anxiety, depression or schizophrenia.
4. Cognitive impairment or mini-mental state examination (MMSE) score ≤24.
5. Severe systemic illness with life-expectancy less than 4 years.
6. Unwillingness to consent for collection of biological samples.
7. Inability to provide informed consent.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Myasthenia Gravis
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-02-08 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Conversion rates from ocular to generalized MG at the last visit and risk factors. | Baseline, 48 months
  Ocular MG patients are followed up to determine the ratio of conversion to generalized disease at the end of follow-up. The clinical records will be retrospectively analyzed to search for risk factors of progressing.
Change in Quantitative Myasthenia Gravis (QMG) Scores from Baseline to 48 months. | Baseline, 12 months, 24 months, 36 months, 48 months
  The QMG is a 13-item scale which measures ocular, bulbar, limb function and respiratory function. The total score ranges from 0 (no myasthenic findings) to 39 (maximal myasthenic deficits) obtained by summing the responses to each individual item (None=0, Mild=1, Moderate=2, Severe=3).
Change in MG-specific Activities of Daily Living scale (MG-ADL). | Baseline,3months, 6 months, 9 months, 12 months, 18 months, 24 months, 30months, 36 months, 42 months, 48 months
  The MG-ADL is an 8-item scale to assess symptoms of myasthenia gravis patients obtained by summing the responses to each individual item (Grades: 0,1,2,3). The score ranges from 0 to 24.
The proportion of patients reaching minimal manifestations (MM) or better. | 48 months
  Clinical statuses of patients are assessed and categorized according to Myasthenia Gravis Foundation of America (MGFA) postintervention status (PIS). MM or better includes Minimal Manifestation (MM), Pharmacologic Remission (PR) or Complete Remission (CR).

SECONDARY OUTCOMES:
Proportion of Patients with Treatment-related Adverse Experiences. | 3 months, 6 months, 12 months, 24 months, 36 months, 48 months
  Treatment-Related Adverse Events (AEs) are evaluated in patients of different regimens.
Changes in titers of MG antibodies. | Baseline, 12 months, 24 months, 36 months, 48 months
  MG antibodies are detected at enrollment and the titers of antibodies will be monitored annually.

CONTACTS AND LOCATIONS:
Overall Officials: yuwei Da, M.D., Study Chair — Xuan Wu Hospital, Capital Medical University
Locations (1):
- Xuan Wu Hospital, Capital Medical University, Beijing, Beijing Municipality, China